CLINICAL TRIAL: NCT06518304
Title: Randomized Controlled Trial: Effectiveness of GentleWave System in Endodontic Treatment and Its Impact on Reducing Post- Operative Pain.
Brief Title: Effectiveness of GentleWave System in Endodontic Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Heilyn Nils, Author- Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1310-8953
Record Dates: First submitted 2024-07-05; First posted 2024-07-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Root Canal Infection; Endodontically Treated Teeth
MeSH Terms: conditions — Pain, Postoperative; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GentleWave (Other): Featuring a handpiece CleanFlow technology, optimizes the delivery of irrigants: initially, a 3% NaOCl solution for 3 or 5 minutes, followed by a water rinse for 15 or 30 seconds, an 8% EDTA solution for 2 minutes, and a final distilled water rinse for 15 or 30 seconds. These solutions penetrate and eliminate necrotic tissue, debris, biofilm and bacteria, leaving the dentin intact and preserving the tooth structure. Use of the Gentlewave system is contraindicated in teeth with immature apices, teeth with insufficient coronal structure, and teeth with root apices that extend into the maxillary sinus.
  Interventions: Other: GentleWave
- Control group (Other): Conventional Syringe Irrigation (CSI), which delivers irrigants (NaOCl, EDTA) through a needle-syringe system. After local anesthesia, the tooth will be isolated with a rubber dam. The pulp chamber will be accessed using ultrasound, eliminating all cavities, restorations with microfiltration or creating access through metal crowns. All canals will be cleaned and shaped with rotary files until at least a canal size of 20.6 or 25.04 is achieved within 0.5 to 1 mm of the apical end. Between each file, 6% NaOCl will be used to disinfect and clean the waste channels. Each canal will then be soaked in 17% EDTA for 1 minute, rinsed with 6% NaOCl, and finally subjected to a final saline rinse. The canals will be filled with root canal sealant and gutta-percha.
  Interventions: Other: Conventional Protocol

INTERVENTIONS:
Other: GentleWave — GentleWave System employs a degassing process that removes dissolved gases from the solution. This optimization prevents the vapor-lock effect and ensures effective energy transmission through the root canal. As the solution enters the pulp chamber, hydrodynamic cavitation occurs, creating microbubbles that implode and generate sound waves across a broad frequency spectrum
  Arms: GentleWave
Other: Conventional Protocol — Delivers irrigants (NaOCl, EDTA) through a needle-syringe system, often fails to reach the entire working length. This inadequacy can result in residual bacteria and necrotic tissue, potentially compromising treatment efficacy and increasing the risk of treatment failure.
  Arms: Control group

SUMMARY:
This study aims to evaluate the efficacy of the GentleWave® System compared to conventional methods in reducing postoperative pain in patients with necrotic pulp or requiring endodontic retreatment.

DETAILED DESCRIPTION:
New irrigation modalities such as the GentleWave® System, which integrates advanced multisonic ultrasound technology, have been developed to overcome limitations and improve root canal treatments success rates, by ensuring comprehensive cleaning while minimizing mechanical instrumentation. This system, featuring CleanFlow technology, optimizes the delivery of irrigants and promotes efficient root canal debridement. Postoperative pain is common, usually peaking within the first 24 hours after treatment and decreasing thereafter.

In the presence of necrosis, microorganisms can colonize anatomical complexities, such as isthmuses, ramifications and dentinal tubules causing symptoms such as pain, inflammation, and in some cases even odontogenic sinusitis. Conventional Syringe Irrigation (CSI), which delivers irrigants (NaOCl, EDTA) through a needle-syringe system, often fails to reach the entire working length and the intricate anatomy of the root canal. This inadequacy can result in residual bacteria and necrotic tissue, potentially compromising treatment efficacy and increasing the risk of treatment failure; furthermore, positive pressure exerted during CSI may cause the extrusion of irrigants beyond the apex, leading to complications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients from 18 years age or older (maximum of 80 years of age), both genders.
* The patients in need of an endodontic intervention.
* All dental groups in both arches were eligible.
* Patients who do or do not experience symptoms after the endodontic intervention.
* Patient-signed informed consent/assent form

Exclusion Criteria:

* Patients< 18 years old.
* fractured teeth.
* Patients who were recommended extraction after the endodontic evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-08-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether using the Gentlewave system demonstrates a significant reduction in the level of postoperative pain after endodontic treatment measured by the VAS (Visual Analog Scale). | 24 hours
  Pain measurements were made using a VAS (Visual Analog Scale of 0-10. Where the value of 0 represented absence of pain and value 10 represented the greatest intensity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- City Endodontics, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No